CLINICAL TRIAL: NCT02375477
Title: Improved Adherence to C. Difficile Isolation Protocols Though Improved Inter-disciplinary Educational Methods
Brief Title: Improved Adherence to C. Difficile Isolation Protocols Through Improved Education Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CASE1815; NCI-2015-00147 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE1815 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Bacterial Infection; Clostridium Difficile
Keywords: Clostridium difficile; C. difficile; adherence
MeSH Terms: conditions — Bacterial Infections | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (isolation protocol education) (Experimental): Residents and nurses are given an educational intervention on isolation protocols for diarrhea and enteric pathogens approved by Infection Control and covering their recommendations.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Given educational presentation
  Other Names: Education for Intervention; Intervention, Educational

SUMMARY:
This clinical trial studies how well inter-disciplinary educational methods work in improving adherence to isolation protocols in patients with Clostridium (C.) difficile infections. An inter-disciplinary educational method may help to prevent the spread of infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To lower rates of C. difficile transmission through improved adherence to recommended isolation protocols.

SECONDARY OBJECTIVES:

I. Improve resident knowledge of infection control procedures and engagement in quality improvement initiatives.

OUTLINE:

Residents and nurses are given a short presentation on isolation protocols for diarrhea and enteric pathogens approved by Infection Control and covering their recommendations.

After completion of study, residents and nurses complete post-tests to determine the effectiveness of the training every 6 months.

ELIGIBILITY:
Patient Criteria

Inclusion Criteria:

* Patient on the gynecologic oncology service
* Admitted to Seidman 6th floor of the Seidman Cancer Center
* Diarrhea or clinical concern for C. difficile infection

Exclusion Criteria:

* None

Medical Staff Criteria:

Inclusion Criteria:

* Any resident or nurse treating a patient meeting the above criteria

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2018-01-06 (Actual)

PRIMARY OUTCOMES:
Rate of C. difficile infection | Up to 1 year
  Rates of infection before vs. after implementation of the intervention will be plotted by quarter and year over the entire study period, to examine possible time trends in the pre-intervention period. Rates during the post-intervention period will be compared to those in the pre-intervention period using logistic regression, adjusting for season of the year, age, race, and other potentially confounding factors.

SECONDARY OUTCOMES:
Proportion of patients with an isolation order placed concurrently with the order for C. difficile | Up to 1 year
  The proportion will be compared pre- vs. post-intervention using logistic regression, adjusting for potentially confounding factors such as season, age, and race. In addition, Kaplan-Meier curves will be used to summarize the time from ordering C. difficile until the isolation order is placed, as well as the time from when the order was placed until it was acknowledged by the nurse, separately for pre- and post-intervention time periods. The curves will be compared between time periods using a logrank or Wilcoxon test allowing for the possibility of censored data.
Difference in scores post-test minus pre-test | Baseline to up to 1 year
  The difference in scores post-test minus pre-test will be calculated for each resident or nurse. The distribution of pre- and post-test scores and of the difference in scores will be summarized graphically and statistically using mean, median, standard deviation, and inter-quartile range. A paired t-test or non-parametric test such as the Wilcoxon signed rank test will be used to test whether there was an improvement in score from pre- to post-test. Analyses will be carried out separately for residents and nurses, as well as for residents and nurses combined.
Retention of information | Up to 1 year
  For residents or nurses who retake the exam, test scores will be summarized graphically and statistically for pre- and post-test, at the original and repeat session. Retention will be gauged by comparing the test score of the re-test with the pre- and post-test scores from the original test, using contrasts in a randomized block analysis of variance model, or using pairwise signed rank tests on the differences in scores.

CONTACTS AND LOCATIONS:
Overall Officials: John Nakayama, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States